CLINICAL TRIAL: NCT01462708
Title: Evaluation of [18F] MK-9470 and PET as a Marker of Cannabinoid-1 Receptor Activity in Subjects With Parkinson Disease Compared With Healthy Controls
Brief Title: Evaluation of [18F]MK-9470 as a Brain Tracer of Cannabinoid-1 Receptor in Parkinson's Disease and Healthy Subjects
Acronym: MK9470
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Danna Jennings, MD, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CB1-01
Record Dates: First submitted 2011-06-08; First posted 2011-10-31 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Molecular NeuroImaging
MeSH Terms: conditions — Parkinson Disease | interventions — MK-9470

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [18F]MK-9470 and PET imaging (Experimental): To Assess [18F]MK-9470 and PET imaging
  Interventions: Drug: [18F]MK-9470

INTERVENTIONS:
Drug: [18F]MK-9470 — Subjects will be injected with 10 mCi, and not to exceed 11 mCi (not >10% of 10 mCi limit)of [18F]MK-9470, followed by PET imaging.
  Other Names: Parkinson Disease; Cannabinoid-1

SUMMARY:
The purpose of this study is to assess MK-9470 Positron Emission Tomography (PET) imaging as a tool to evaluate the activity of the CB-1 receptor in the brain.

DETAILED DESCRIPTION:
The underlying goal of this study is to assess MK-9470 PET imaging as a tool to evaluate the activity of the CB-1 receptor in the brain of Parkinson's Disease (PD) research participants.

ELIGIBILITY:
Early PD Subjects

Inclusion criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a diagnosis of PD (based on UK Brain Bank Criteria) within the past 2 years.
* Modified Hoehn and Yahr stages 1-2.
* No evidence of dyskinesia by history or clinical examination
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-MK-9470 injection.

Advanced PD subjects

Inclusion criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a diagnosis of PD (based on UK Brain Bank Criteria) of at least 5 years duration.
* Modified Hoehn and Yahr stages 1-4.
* No evidence of dyskinesia by history or clinical examination
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-MK-9470 injection.

Subjects who have a clinical diagnosis of advanced PD with dyskinesia will be recruited for this study.

ePD subjects

Inclusion criteria:

* The participant is 30 years or older.
* Written informed consent is obtained.
* Participants have a diagnosis of PD (based on UK Brain Bank Criteria) of at least 5 years.
* Modified Hoehn and Yahr stages 1-4.
* Evidence of dyskinesia either by history or clinical examination
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-MK-9470 injection.

PD (all stages- e-PD, aPD, aPD-dys)Subject Selection. Subjects who have a clinical diagnosis of ePD, aPD, aPD-dys will be recruited for this study.

All PD subjects

Exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The patient has evidence of unstable gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, pulmonary, or other disorder or disease.
* Evidence of a stroke or mass lesion in a clinically relevant area that may interfere with the imaging outcome measure
* Subjects with radiation exposure above acceptable levels
* Pregnancy

Healthy Control Subject Selection: subjects who have no neurological disease will be recruited for this study.

Healthy control subjects

Inclusion criteria:

* The participant is 18 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F]-MK9470 injection.

Exclusion criteria:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* Subjects with radiation exposure above acceptable levels
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Dynamic uptake and washout of [18F]MK-9470 | Approximately 2 years
  To assess the dynamic uptake and washout of [18F]-MK-9470 in brain using positron emission tomography (PET) in early Parkinson disease and advanced Parkinson disease with and without dyskinesia and similarly aged healthy control subjects as a potential imaging biomarker of the cannabionoid-1 (CB-1) receptor in brain.

SECONDARY OUTCOMES:
To acquire safety data | Approximately 2 years
  Safety will be assessed by the number of adverse events experienced by subjects and any clinically significant changes in laboratory tests or vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- See also: Institute for Neurodegenerative Disorders — http://www.indd.org